CLINICAL TRIAL: NCT06758336
Title: Caffeinated Chewing Gum Improves Sympathetic Nerve Activity and Simulates Wrestling Performance: a Double-blind Crossover Trial
Brief Title: Caffeinated Chewing Gum & Wrestling Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113-9
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Caffeine; Control
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: a randomized crossover double-blind study design
Who Masked: Participant, Investigator
Masking Description: placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine gum (Experimental): The participants chewing caffeine gum 10 minutes before exercise
  Interventions: Dietary Supplement: caffeine
- placebo gum (Placebo Comparator): The participants chewing placebo gum 10 minutes before exercise
  Interventions: Dietary Supplement: caffeine

INTERVENTIONS:
Dietary Supplement: caffeine — The participants chewing either caffeine Gum (CAF trial, containing 3 mg/kg of caffeine) for 10 minutes. After rested for 15 minutes, the participants underwent tests.

SUMMARY:
The purpose of this study was to investigate the effect of caffeinated chewing gum on sympathetic nerve activity on wrestling simulation match.

DETAILED DESCRIPTION:
The purpose of this study was to investigated whether caffeine intake is effective in improving the performance of wrestlers in a simulated competition. The study was designed to involve 16 healthy adult male athletes who had been trained in professional wrestling and were divided into caffeine trial (CAF trial) and placebo trial (PL trial) in a randomized crossover double-blind study design. After three days of dietary control, participants arrived at the laboratory in the afternoon of the day of the trial to collect saliva samples in a quiet state and were fitted with a heart rate monitor. Participants chewed either caffeine-containing gum at 3 mg/kg body weight (CAF trial) or placebo-containing gum without caffeine (PL trial) for 10 minutes and then spit it out. Participants then underwent a 15-minute dynamic warm-up. At the end of the warm-up, participants performed 2 rounds of 3-minute wrestling-specific simulated matches, and the number of falls in the simulated matches was recorded. After the simulation match, saliva samples were collected from the participants again. The saliva samples were analyzed for caffeine alpha-amylase concentration. Differences between the two trials were analyzed using a paired sample t-test and significance was set at α<0.05.

ELIGIBILITY:
Inclusion Criteria:

* more than 6years of professional wrestling training;
* more than 6 months of continuous training;
* recovering from sports injuries such as strains and contusions for at least 3 months.

Exclusion Criteria:

* non-professionally wrestling athlete;
* none regular training in the past 6 months;
* less than 3 months of recovery from a sports injury, or present epilepsy, hypertension, hyperlipidemia, heart disease, arthritis, osteoporosis, or brain injury;
* a history of caffeine allergy.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male
Enrollment: 16 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
The number of falls in the simulated matches | 15 minutes after intervention
  Record number of falls in the simulated matches

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hui Chiu, PhD, Principal Investigator — Sport Science Research Center
Locations (1):
- National Taiwan University of Sport, Taichung, North, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan

DOCUMENTS (1):
  • Study Protocol (2024-12-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT06758336/Prot_000.pdf